CLINICAL TRIAL: NCT01441739
Title: Intestinal Failure in Necrotising Enterocolitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 04-197
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- NEC suspected - Final diagnosis NEC
- NEC suspected - Final diagnosis no NEC
- Controls

SUMMARY:
Necrotizing enterocolitis (NEC) is a severe gastrointestinal disorder with high morbidity and mortality (20-40%), affecting predominantly premature neonates. NEC continues to present a diagnostic challenge to clinicians. The initial clinical manifestations of NEC are non-specific and indistinguishable from other gastrointestinal disorders and sepsis.

The first goal of this study is to find and evaluate tests to diagnose NEC at an early stage. For the development of new diagnostic markers, the investigators require knowledge of pathophysiological processes that underlie NEC, which still remain unclear. Therefore, the second goal of this study is to elucidate the etiology of NEC. Furthermore, understanding of the pathophysiology of NEC can offer the possibility to develop new therapeutical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with abdominal signs suspected of NEC
* All neonates admitted to the NICU of the Maastricht University Medical Center between July 2007 and July 2008

Exclusion Criteria:

* No written informed consent of both parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates with abdominal signs suspected of NEC All neonates admitted to the NICU of the Maastricht University Medical Center between July 2007 and July 2008
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2004-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Urinary I-FABP | Within the first 30 days (plus or minus 3 days) after clinical suspicion of NEC

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - University Medical Center Utrecht, Utrecht